CLINICAL TRIAL: NCT04101487
Title: A Cluster Randomized Trial to Study the Effect of Cash Transfers and Nutrition Education on Dietary Diversity Among Children 6-23 Months of Age in Grand Gedeh County, Liberia: a Pilot Study
Brief Title: Cash Transfers to Increase Dietary Diversity in Grand Gedeh County, Liberia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Michelle Niescierenko, Assistant Professor of Pediatrics and Emergency Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00031767
Record Dates: First submitted 2019-06-27; First posted 2019-09-24 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2023-03

CONDITIONS: Malnutrition, Child
Keywords: Cash Transfers; Liberia; Stunting; Dietary diversity
MeSH Terms: conditions — Child Nutrition Disorders; Growth Disorders | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Participants in this arm will receive routine monthly visits along with survey administration and the regular package of health services provided at the facility level and at home by community health assistants
- Cash Transfers (Experimental): Participants in this arm will receive routine monthly visits along with the regular package of health services provided at the facility level and at home by community health assistants and unconditional cash transfers every month
  Interventions: Other: Cash Transfer
- Cash Transfers and Nutrition Education (Experimental): Participants in this arm will receive routine monthly visits along with the regular package of health services provided at the facility level and at home by community health assistants, unconditional cash transfers every month, and structured nutrition education provided at household level by community health assistants based on a structured nutrition education handbook.
  Interventions: Other: Cash Transfers and Nutrition Education

INTERVENTIONS:
Other: Cash Transfer — Monthly cash transfers
  Arms: Cash Transfers
Other: Cash Transfers and Nutrition Education — Cash transfers every month and structured nutrition education provided at household level by community health assistants based on a nutrition education handbook
  Arms: Cash Transfers and Nutrition Education

SUMMARY:
The investigators aim to evaluate the efficacy of a cash transfer and nutrition education program delivered by community health assistants to increase dietary diversity among children 6 to 23 months of age in Grand Gedeh County, Liberia.

DETAILED DESCRIPTION:
Worldwide, more than one in five children suffer from chronic malnutrition. In Liberia, there are more than 230,000 children suffering from chronic malnutrition and 32% of children under five are stunted. Previous studies have shown that inadequate dietary diversity is strongly associated with stunting in children under two years of age. An interventional package including cash transfers and education has the potential to improve dietary diversity and long-term outcomes such as improved growth and reduced rates of stunting among children.

The investigators' objective is to evaluate the efficacy of a cash transfer and nutrition education program delivered by community health assistants to increase dietary diversity among children 6 to 23 months of age in Grand Gedeh County, Liberia. The investigators will conduct a pilot, cluster randomized trial in 45 communities. The investigators hypothesize that a multi-pronged interventional package aimed at strengthening the household environment will result in improved dietary diversity for children 6 to 23 months of age. Moreover, the investigators also hypothesize that unconditional cash transfers will result in improved dietary diversity for children 6 to 23 months of age in Grand Gedeh County, Liberia.

ELIGIBILITY:
Inclusion Criteria:

* Participants 6 to 23 months of age
* Participants with consenting caregivers to have monthly visits and to participate in the program
* Caregivers of all ages will be included

Exclusion Criteria:

* Participants who are younger than 6 months of age (children < 6 months of age are encouraged to exclusively breastfeed, making dietary diversity irrelevant in this age group)
* Participants older than 23 months of age
* Participants with non-consenting caregivers

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 599 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in proportion of children 6 to 23 months of age who meet minimum dietary diversity scores (DDS) over the study period as reported by caregivers | 6 months
  The DDS has been widely used to measure the sum of diverse food groups consumed in a 24-hour period

SECONDARY OUTCOMES:
Meal frequency | 6 months
  Mean self-reported meal frequency over the 24-hour period prior to monthly CHA visits
Increase in child weight in kilograms | 6 months
  changes in child weight in kilograms during the study period measured with digital scale (UNISCALE)
Increase in mid upper arm circumference in centimeters | 6 months
  changes in mid upper arm circumference in centimeters measured with MUAC tape measure
Increase in child length/height in centimeters | 6 months
  changes in child length/height in centimeters during the study period measured with Height Board
Health care utilization (clinic) | 6 months
  number of clinic visits for illnesses (including type of illness)
Health care utilization (hospital) | 6 months
  hospitalizations (if any) during the study period
Health care utilization (antimicrobials) | 6 months
  use of antibiotics/antimalarials during the study period
Health care utilization (nutritional support) | 6 months
  if the child received supplementary nutritional support (e.g. ready to use therapeutic food RUTF)
Knowledge, attitudes, and practices | 6 months
  caregiver's knowledge, attitudes, and practices (KAP) of infant and young child feeding

CONTACTS AND LOCATIONS:
Locations (1):
- Grand Geddeh County Health Office, Zwedru, Liberia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rees CA, Cleon D, Davis AB, Sammy AM, Britto CD, Massaquoi W, Forkpa OW, Johnson AJ, Hook VF, MaCauley JA, Pewu GF, Gorpue M, Gborie A, Brown TT, Fannieh A, Dweh T, Marley RB, Baysah MK, Nowine NN, Niescierenko M, Zaizay L. Cash transfers and nutrition education to improve dietary diversity among children aged 6-23 months in Grand Gedeh County, Liberia: a cluster-randomized trial. J Trop Pediatr. 2022 Oct 6;68(6):fmac096. doi: 10.1093/tropej/fmac096. PMID 36350714